CLINICAL TRIAL: NCT04160325
Title: The Effect of the Exclusive Enteral Nutrition Combined With Azathioprine in Maintaining Remission of Patients With Crohn's Diseases After Surgery
Brief Title: Effect of the Exclusive Enteral Nutrition Combined With Azathioprine for Remission of Crohn's Diseases After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhu Weiming (Other)
Responsible Party: Sponsor-Investigator, Zhu Weiming, Director, Head of General Surgery, Principal Investigator, Clinical Professor, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: jinlingH201709
Record Dates: First submitted 2019-11-03; First posted 2019-11-13 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Postoperative Period; Azathioprine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 months exclusive enteral nutrition plus azathioprine (Experimental): patients underwent surgery in this arm will given 3 months exclusive enteral nutrition,and free diet after 3 months. All patients will be adminsrated with oral azathioprine to preventing disease recurrence.
  Interventions: Dietary Supplement: postoperative 3-month exclusive enteral nutrition; Drug: azathioprine
- normal diet plus azathioprine (Active Comparator): patients underwent surgery in this arm will given free diet all through. All patients will be adminsrated with oral azathioprine to preventing disease recurrence.
  Interventions: Drug: azathioprine; Other: normal diet

INTERVENTIONS:
Dietary Supplement: postoperative 3-month exclusive enteral nutrition — postoperative 3-month exclusive enteral nutrition after surgery and alter to normal food after 3 months
  Arms: 3 months exclusive enteral nutrition plus azathioprine
Drug: azathioprine — azathioprine
Other: normal diet — normal diet
  Arms: normal diet plus azathioprine

SUMMARY:
for some patients with Crohn's diseases undergoing surgery，whether exclusive enteral nutrition(EEN) could delay the disease relapse needs exploration.The trial will study whether the efficacy of postoperative EEN could help keeping remission.

DETAILED DESCRIPTION:
For patients with Crohn's disease(CD), whether exclusive enteral nutrition(EEN) following bowel resection and anastomosis could delay the disease recurrence remains unkown. In this study， CD patients after surgery will be divided into two groups: one group is treated with 3 months' EEN and then turn to normal diet after 3 months; the other group is given with normal diet all through. All patients will be adminstrated with oral azathioprine after surgery. Then, the rates of 1 year postoperative endoscopic recurrence will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* CD patients who undergoing bowel resection with anastomosis

Exclusion Criteria:

* patients who had administered with immunomodulators or biological agents patients who were created stoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
the 1 year postoperative anastomotic recurrence | 1 year
  the 1 year postoperative anastomotic recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Jinling hosptal,Medical School of Nanjing University, Nanjing, Jiangsu, China